CLINICAL TRIAL: NCT00784316
Title: Intravenous Metoprolol Versus Intravenous Amiodarone in the Prevention of Atrial Fibrillation After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Tampere University Hospital (Other); Vaasa Central Hospital, Vaasa, Finland (Other)
Responsible Party: Principal Investigator, Jari Halonen, MD,PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KUH5204005
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Atrial Fibrillation; Cardiac Surgery
Keywords: Prevention
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metoprolol; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metoprolol (Active Comparator)
  Interventions: Drug: metoprolol, amiodarone
- amiodarone (Active Comparator)
  Interventions: Drug: metoprolol, amiodarone

INTERVENTIONS:
Drug: metoprolol, amiodarone — to compare the effectiviness of intravenous administration of metoprolol and amiodarone in the prevention of atrial fibrillation after cardiac surgery

SUMMARY:
The aim of the study is to test the efficiency of intravenous administration of metoprolol versus intravenous administration of amiodarone in the prevention of atrial fibrillation after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective CABG and aortic valve patients in cardiac surgery,
* previous use of betablocker therapy

Exclusion Criteria:

* previous atrial fibrillation or flutter,
* thyroid disease,
* uncontrolled heart failure,
* II or III degree atrioventricular block

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Halonen jari, Kuopio, Finland

REFERENCES:
- [Derived] Halonen J, Loponen P, Jarvinen O, Karjalainen J, Parviainen I, Halonen P, Magga J, Turpeinen A, Hippelainen M, Hartikainen J, Hakala T. Metoprolol versus amiodarone in the prevention of atrial fibrillation after cardiac surgery: a randomized trial. Ann Intern Med. 2010 Dec 7;153(11):703-9. doi: 10.7326/0003-4819-153-11-201012070-00003. PMID 21135293